CLINICAL TRIAL: NCT03683134
Title: A Pilot, Theory-Based, Nutrition Intervention Promoting a Mediterranean Diet for the Reduction of Cardiovascular Disease Risk Factors in a High-Risk Population of the Southeastern United States: The Healthy Hearts Program (HHP)
Brief Title: A Mediterranean Diet Nutrition Education Program for the Reduction of Cardiovascular Disease Risk in the Southeastern U.S.
Acronym: HHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Michael W. Greene, Director, Auburn University Metabolic Phenotyping Laboratory, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: The Healthy Hearts Program
Record Dates: First submitted 2018-09-20; First posted 2018-09-25 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Obesity
Keywords: Cardiovascular Disease; Mediterranean Diet; Nutrition education
MeSH Terms: conditions — Cardiovascular Diseases; Obesity | interventions — Diet, Mediterranean; Olive Oil; American Heart Association

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet group (Experimental): Participants will receive both nutrition education on patterns of a Mediterranean style diet as well as olive oil and mixed nuts.
  Interventions: Behavioral: Mediterranean diet; Dietary Supplement: Olive oil and mixed nuts
- American Heart Association group (Active Comparator): Participants will receive nutrition education on the dietary recommendations for heart health from the American Heart Association.
  Interventions: Behavioral: American Heart Association

INTERVENTIONS:
Behavioral: Mediterranean diet — Participants will receive nutrition education and educational materials from a registered dietitian on patients on the patterns of a Mediterranean style diet. Seven education sessions will be delivered through an online platform. Participants will be asked to complete one education session per week for the first six weeks and the final session at week 9.
  Arms: Mediterranean diet group
Dietary Supplement: Olive oil and mixed nuts — Participants in the Mediterranean diet group will receive 3 liters of extra-virgin olive oil and 3 pounds of mixed nuts (1.5 pounds raw almonds and 1.5 pounds raw walnuts) at baseline and at 6 weeks. Participants will be educated by oral and written means, on consumption goals of the nuts and olive oil.
  Arms: Mediterranean diet group
Behavioral: American Heart Association — Participants will receive nutrition education and educational materials from a registered dietitian on patients on the dietary recommendations from the American Heart Association for heart health. Seven education sessions will be delivered through an online platform. Participants will be asked to complete one education session per week for the first six weeks and the final session at week 9.
  Arms: American Heart Association group

SUMMARY:
A 12-week, randomized nutrition intervention for the reduction of cardiovascular disease risk factors in a high-risk population in the southeastern United States. The primary objective of this pilot study was to assess the efficacy of a Mediterranean diet intervention (education + extra-virgin olive oil (EVOO) and mixed nut supplementation) versus that of an American Heart Association (AHA) nutrition intervention (education) on serum blood lipid levels as markers for cardiovascular disease risk. Researchers conducting this trial hypothesize that a greater reduction will be seen in cardiovascular disease risk factors in the Mediterranean diet intervention.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Auburn University's health insurance program during the course of the study or a dependent of the enrollee during the course of the study
* BMI >24.9 (kg/m2)
* AND Meets two or more of the following
* Screening values classified in the "yellow" or "red" zone for:
* Systolic blood pressure (mmHg): Yellow zone: ≥140, Red zone: ≥160;
* Diastolic Blood pressure (mmHg): Yellow zone: ≥90, Red zone: ≥ 100;
* Fasting blood glucose (mm/dL): Yellow zone: ≥100, Red zone: ≥ 126
* Blood glucose (random) (mg/dL): Yellow zone: 140-200, Red zone > 200
* Total Cholesterol (mg/dL): Yellow zone: ≥200, red zone: ≥250
* Have a pre-existing diagnosis of hypertension, pre-diabetes, or hypercholesterolemia
* Current smoker (≥1 cigarette/day)
* Are: male (age: 55-80) or female (age: 60-80)
* A family history of premature coronary heart disease
* High risk ethnicity: Black, African American, American Indians/Alaska Natives, Non-Hispanic blacks, Mexican-Americans, Asian, Hispanic/Latino

Exclusion Criteria:

* Minors that are less than 19 years of age
* Individuals who are not enrolled in the Auburn University health insurance program for the 2016 plan year at baseline and have not yet completed initial visit
* Individuals who have not completed their 2015 "Healthy Tigers" biometric screening between January 1st and December 31st, 2015 (these can be completed by the "Healthy Tigers" staff or by submitting a healthcare provider form from the individuals' physician to the "Healthy Tigers" office), unless enrolled in "TigerMeds".
* Individuals who are pregnant or who intend to become pregnant during the 12-week health and wellness challenge.
* Individuals who anticipate absence or travel throughout the study that would interfere with their ability to complete the analysis at the mid-point and end of challenge.
* Patients with a peanut, tree nut, or olive oil food allergy or intolerance.
* Patients who are unable or unwilling to travel to Auburn University main campus for live health and wellness challenge events, individual assessments, personal appointments, and pre- and post- data collection
* Individuals who have NOT been stabilized on medication to treat or manage high blood pressure, high cholesterol, dyslipidemia, or pre diabetes for at least 12 weeks prior to the study.
* Patients who do not have access to the internet and therefore unable to complete the education portion of the study
* Individuals who have a pacemaker
* Patients who decline participation during informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure Measurement | Change from at baseline blood pressure to 6-weeks
  Measured in mmHg
Systolic Blood Pressure Measurement | Change from at baseline blood pressure to 12-weeks
  Measured in mmHg

SECONDARY OUTCOMES:
Diastolic Blood Pressure Measurement | Change from at baseline weight to 6-weeks
  Measured in mmHg
Change in Weight | Change from at baseline weight to 12-weeks
  Measured in kilograms (kg)
Calculation of Body Mass Index (BMI) (kg/m∧2) | Change from baseline weight to 6-weeks
  Height in meters will be combined with weight in kilograms will be combined to report BMI in kg/m∧2)
Calculation of BMI (kg/m∧2) | Change from baseline weight to 12-weeks
  Height in meters will be combined with weight in kilograms will be combined to report BMI in kg/m∧2)
Concentration of fasted total cholesterol | Change from baseline weight to 6-weeks
  Measured in mg/dL
Concentration of fasted total cholesterol | Change from baseline weight to 12-weeks
  Measured in mg/dL
Concentration of fasted high-density lipoprotein (HDL) cholesterol | Change from baseline weight to 6-weeks
  Measured in mg/dL
Concentration of fasted high-density lipoprotein (HDL) cholesterol | Change from baseline weight to 12-weeks
  Measured in mg/dL
Concentration of fasted low-density lipoprotein (LDL) cholesterol | Change from baseline weight to 12-weeks
  Measured in mg/dL
Concentration of fasted low-density lipoprotein (LDL) cholesterol | Change from baseline weight to 6-weeks
  Measured in mg/dL
Concentration of fasted triglycerides | Change from baseline weight to 6-weeks
  Measured in mg/dL
Concentration of fasted triglycerides | Change from baseline weight to 12-weeks
  Measured in mg/dL
A calculation of total cholesterol (mg/dL) to HDL (mg/dL) ratio | Change from baseline weight to 12-weeks
  Total cholesterol (mg/dL) will be used with HDL (mg/dL) to calculate total cholesterol to HDL ratio
A calculation of total cholesterol (mg/dL) to HDL (mg/dL) ratio | Change from baseline weight to 6-weeks
  Total cholesterol (mg/dL) will be used with HDL (mg/dL) to calculate total cholesterol to HDL ratio
Concentration of fasted blood glucose | Change from baseline weight to 6-weeks
  Measured in mg/dL
Concentration of fasted blood glucose | Change from baseline weight to 12-weeks
  Measured in mg/dL
A calculation of waist (inches) to height (inches) ratio | Change from baseline weight to 12-weeks
  Waist circumference in inches will be calculated with height measurement in inches to report the waist-to-height ratio
A calculation of waist (inches) to height (inches) ratio | Change from baseline weight to 6-weeks
  Waist circumference in inches will be calculated with height measurement in inches to report the waist-to-height ratio
Calculation of homeostatic model assessment (HOMA)-insulin resistance (IR) from fasted blood concentrations of fasted blood glucose and fasted insulin | Change from baseline weight to 6-weeks
  Fasting plasma glucose in mg/dL and fasting serum insulin in milliUnits (mU)/I will be used to calculate HOMA-IR as an indicator for insulin resistance.
Calculation of homeostatic model assessment (HOMA)-insulin resistance (IR) from fasted blood concentrations of fasted blood glucose and fasted insulin | Change from baseline weight to 12-weeks
  Fasting plasma glucose in mg/dL and fasting serum insulin in mU/I will be used to calculate HOMA-IR as an indicator for insulin resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Greene, PhD, Study Chair — Auburn University; Amy W Willis, MS, RD, Principal Investigator — Auburn University
Locations (1):
- Auburn University Pharmaceutical Care Center, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT03683134/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT03683134/ICF_001.pdf